CLINICAL TRIAL: NCT00001758
Title: Continued Salvage Anti-Retroviral Therapy With Abacavir, Amprenavir, and Efavirenz
Brief Title: Continued Antiretroviral Therapy With Abacavir, Amprenavir and Efavirenz
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980031; 98-I-0031
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: HIV Infection
Keywords: Antiretroviral; HIV-1; 1592U89; 141W94; DMP 266
MeSH Terms: conditions — HIV Infections | interventions — abacavir; amprenavir; efavirenz

INTERVENTIONS:
Drug: Abacavir
Drug: Amprenavir
Drug: Efavirenz

SUMMARY:
This study will continue to treat and collect safety and efficacy data on patients who participated in Glaxo-Wellcome's multi-center study on combination therapy with abacavir, amprenavir and efavirenz (A Phase II Study Evaluating the Safety and Antiviral Activity of Combination Therapy with 1592U89, 141W94 and DMP 266 (Sustiva) in HIV-1 Infected Subjects with Detectable [greater than 400 Copies/mL] HIV-1 Plasma RNA Despite Treatment with a Protease Inhibitor-Containing Regimen).

HIV-infected patients 18 years of age and older who participated in the above study at the NIH site may be eligible for the current study. Participants will be followed every 3 months with a general health evaluation and laboratory tests. This is a NIH study, and information will not be provided to Glaxo Wellcome

DETAILED DESCRIPTION:
In this open-label, single-arm study, HIV-1 infected patients who had, at study entry, a viral burden of at least 500 copies/mL despite 20 weeks of treatment with a protease inhibitor receive combination therapy with three antiretroviral agents that were investigational at the start of study but have since been approved: abacavir, amprenavir, and efavirenz. At the end of 16 weeks, the addition of other antiretroviral agents to the study regimen was permitted. This was originally a multi-center study, but it has been closed at all other sites. It remains open at the NIH to continue to provide therapy to subjects who have received benefit as determined by a decline in viral load from baseline. Safety and viral load data continue to be collected.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA:

Subjects who were previously enrolled in this protocol when it was a multi-center study and who signed the new informed consent were enrolled. There has been and will be no other new enrollment. Thus, subjects who were not previously enrolled are excluded.

Subjects are adults infected with HIV-1 who had, prior to study enrollment, a plasma viral load of at least 500 copies/mL despite at least 20 weeks of treatment with a protease inhibitor and without change in protease inhibitor therapy in the 12 weeks prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1997-11; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Livington DJ, Pazhanisamy S, Porter DJ, Partaledis JA, Tung RD, Painter GR. Weak binding of VX-478 to human plasma proteins and implications for anti-human immunodeficiency virus therapy. J Infect Dis. 1995 Nov;172(5):1238-45. doi: 10.1093/infdis/172.5.1238. PMID 7594659
- [Background] Partaledis JA, Yamaguchi K, Tisdale M, Blair EE, Falcione C, Maschera B, Myers RE, Pazhanisamy S, Futer O, Cullinan AB, et al. In vitro selection and characterization of human immunodeficiency virus type 1 (HIV-1) isolates with reduced sensitivity to hydroxyethylamino sulfonamide inhibitors of HIV-1 aspartyl protease. J Virol. 1995 Sep;69(9):5228-35. doi: 10.1128/JVI.69.9.5228-5235.1995. PMID 7636964
- [Background] Tisdale M, Myers RE, Maschera B, Parry NR, Oliver NM, Blair ED. Cross-resistance analysis of human immunodeficiency virus type 1 variants individually selected for resistance to five different protease inhibitors. Antimicrob Agents Chemother. 1995 Aug;39(8):1704-10. doi: 10.1128/AAC.39.8.1704. PMID 7486905